CLINICAL TRIAL: NCT07233668
Title: Immediate Versus Deferred Cytoreductive Nephrectomy With Ipilimumab/Nivolumab in Metastatic Clear Cell Renal Cell Carcinoma: A Multicenter, Randomized, Open-Label, Phase III Trial
Brief Title: Immediate Versus Deferred Cytoreductive Nephrectomy With Ipilimumab/Nivolumab in mRCC
Acronym: IVE in mRCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang Wook Jeong, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2502-014-1611
Record Dates: First submitted 2025-09-03; First posted 2025-11-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Renal Cell Carcinoma ( mRCC)
Keywords: Metastatic Renal Cell Carcinoma; Immune Checkpoint Inhibitor; Cytoreductive Nephrectomy; Progression-Free Survival; Randomized Clinical Trial
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront Cytoreductive Nephrectomy (CN) (Experimental): Participants will undergo immediate cytoreductive nephrectomy. About 4 weeks after surgery, they will receive induction therapy with ipilimumab plus nivolumab for 4 cycles, followed by maintenance nivolumab. Regular assessments of progression, perioperative complications, safety, and quality of life will be performed for 15 months.
  Interventions: Drug: Ipilimumab plus Nivolumab; Procedure: Cytoreductive Nephrectomy
- Deferred Cytoreductive Nephrectomy (CN) (Experimental): Participants will first receive 4 cycles of ipilimumab plus nivolumab induction therapy. After reassessment, they will undergo deferred cytoreductive nephrectomy, followed by maintenance nivolumab. Safety, perioperative complications, progression, and quality of life will be evaluated regularly for 15 months
  Interventions: Drug: Ipilimumab plus Nivolumab; Procedure: Cytoreductive Nephrectomy

INTERVENTIONS:
Drug: Ipilimumab plus Nivolumab — Participants will receive 4 cycles of ipilimumab combined with nivolumab as induction therapy, followed by nivolumab maintenance depending on randomization schedule (before or after surgery).
Procedure: Cytoreductive Nephrectomy — Surgical removal of the primary kidney tumor (cytoreductive nephrectomy), performed either upfront (before systemic therapy) or deferred (after 4 cycles of ipilimumab/nivolumab induction), depending on randomization arm.

SUMMARY:
The goal of this clinical trial is to learn whether the timing of surgery (cytoreductive nephrectomy) improves outcomes when combined with immunotherapy (ipilimumab and nivolumab) in adults with metastatic clear cell renal cell carcinoma.

The main questions this study aims to answer are:

* Does upfront (immediate) surgery before immunotherapy improve survival compared to delayed surgery after immunotherapy?
* What medical problems (side effects or complications) occur with each treatment sequence?
* How do the two strategies affect quality of life?

Researchers will compare two groups:

* Upfront surgery group: Participants will have surgery first, then receive 4 cycles of ipilimumab/nivolumab, followed by nivolumab maintenance.
* Deferred surgery group: Participants will receive 4 cycles of ipilimumab/nivolumab first, then surgery, followed by nivolumab maintenance.

Participants will:

* Be randomly assigned to one of the two groups
* Undergo regular clinic visits, imaging tests, and blood collections for safety and biomarker studies
* Be followed for 15 months to check disease progression, complications, survival, and quality of life

This trial will help determine the best timing for surgery in the era of immunotherapy and provide evidence for improved treatment strategies for patients with metastatic kidney cancer

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label phase III trial designed to evaluate the optimal timing of cytoreductive nephrectomy (CN) in patients with synchronous metastatic clear cell renal cell carcinoma (mRCC) in the era of immune checkpoint inhibitors.

Although CN has historically been considered standard in mRCC, the timing of surgery (immediate vs deferred) remains controversial, particularly after the introduction of immune checkpoint blockade. Recent retrospective studies and meta-analyses suggest potential survival benefits of deferred CN following systemic therapy, but high-level prospective evidence is lacking.

In this study, participants with intermediate or poor IMDC risk mRCC will be randomized into two groups:

* Upfront CN arm: Patients undergo immediate CN followed by 4 cycles of ipilimumab plus nivolumab (Ipi/Nivo) and then nivolumab maintenance.
* Deferred CN arm: Patients receive 4 cycles of Ipi/Nivo induction first, followed by CN, and then nivolumab maintenance.

The primary endpoint is progression-free survival (PFS). Secondary endpoints include overall survival (OS), perioperative morbidity, radiologic response, rate of unresectable tumors in the deferred group, impact of CN on early progression, surgical outcomes, and quality of life. Exploratory endpoints include biomarker studies using peripheral blood mononuclear cells (PBMCs) to characterize responders vs non-responders to Ipi/Nivo.

Patients will be followed for 15 months after treatment initiation, with regular imaging, clinical assessments, and laboratory monitoring. Approximately 172 patients across 12 institutions in Korea will be enrolled.

The results of this trial are expected to establish high-level evidence regarding the role and optimal timing of CN in mRCC, improve clinical decision-making, and provide guidance for treatment strategies in the immuno-oncology era

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all of the following:
* Age ≥ 19 years (male or female).
* Histologically confirmed synchronous metastatic clear cell renal cell carcinoma.
* ECOG performance status 0-1.
* At least one measurable metastatic lesion (per RECIST v1.1).
* Primary renal tumor considered surgically resectable.
* IMDC intermediate- or poor-risk classification.
* Estimated life expectancy > 3 months.
* Ability to understand and voluntarily sign informed consent.

Exclusion Criteria:

* Prior systemic therapy for metastatic RCC.
* History of another malignancy diagnosed or treated within 2 years (except for cured non-melanoma skin cancer or in-situ cancers).
* Significant comorbid conditions making participation inappropriate, such as:

Moderate to severe cardiovascular, cerebrovascular, pulmonary, or hepatic disease.

* History or suspicion of autoimmune disease incompatible with immune checkpoint inhibitor therapy.
* Requirement for systemic corticosteroid therapy >10 mg/day prednisone equivalent, or other immunosuppressive drugs.
* Any other condition judged by the investigator to make the patient unsuitable for trial participation.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) assessed by RECIST version 1.1 | Up to 15 months after treatment initiation
  Time from randomization to first documented disease progression or death from any cause, whichever occurs first. Disease progression will be assessed according to RECIST version 1.1 criteria and clinical evaluation.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 15 months after treatment initiation
  Time from randomization to death from any cause.
Rate and Severity of Perioperative Complications Assessed by Clavien-Dindo Classification | Within 90 days after cytoreductive nephrectomy
  Proportion of patients experiencing perioperative complications graded using the Clavien-Dindo classification (Grades I-V).
Rate and Severity of Perioperative Adverse Events Assessed by CTCAE v4.0 | Within 90 days after cytoreductive nephrectomy
  Severity of postoperative adverse events graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Grade 1-5).
Radiologic Tumor Response Rate Assessed by RECIST v1.1 | At baseline, at 12 weeks (after 4 cycles of ipilimumab/nivolumab induction therapy), and every 12 weeks thereafter up to 15 months
  Rate of complete response (CR) and partial response (PR) to ipilimumab/nivolumab, assessed using RECIST version 1.1.
Rate of Unresectable Tumors in the Deferred Arm | At the time of planned deferred cytoreductive nephrectomy
  Proportion of participants in the deferred arm with tumors deemed unresectable at surgery.
Early Disease Progression Rate Within 4 Weeks Post-Nephrectomy | Within 4 weeks of cytoreductive nephrectomy
  Proportion of patients showing disease progression (PD) within 4 weeks after surgery in both arms.
Rate of Open vs Minimally Invasive Surgical Approach | At time of cytoreductive nephrectomy
  Proportion of surgeries performed using open or minimally invasive techniques.
Extent of Surgery (e.g., Radical vs Partial Nephrectomy; Lymphadenectomy Yes/No) | At time of cytoreductive nephrectomy
  Surgical extent categories documented at time of surgery.
Quality of Life Assessed by FACT-Kidney Symptom Index 15-item (FKSI-15) | Baseline, at 12 weeks (after 4 cycles of therapy), and every 12 weeks thereafter up to 15 months
  Quality of life measured using the Functional Assessment of Cancer Therapy - Kidney Symptom Index 15-item (FKSI-15) questionnaire.
  The total score ranges from 0 to 60, with higher scores indicating better quality of life and fewer kidney cancer-related symptoms.
Quality of Life Assessed by EORTC QLQ-C30 | Baseline, at 12 weeks (after 4 cycles of therapy), and every 12 weeks thereafter up to 15 months
  Patient-reported outcomes evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). Scores for each domain range from 0 to 100.
Health Utility Score Assessed by EQ-5D-5L | Baseline, at 12 weeks (after 4 cycles of therapy), and every 12 weeks thereafter up to 15 months
  Health status measured using the EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire.
  The EQ-5D-5L utility index score typically ranges from <0 (health states worse than death) to 1 (full health), with higher scores representing better overall health status.
  The EQ-VAS records self-rated health on a 0-100 scale, where higher scores indicate better perceived health.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, MD, PhD, Principal Investigator — Seoul National Universtiy Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant-level data will not be shared due to privacy concerns and local regulations. Only aggregate study results will be published in peer-reviewed journals and scientific meetings.

REFERENCES:
- [Background] Esagian SM, Karam JA, Msaouel P, Makrakis D. Upfront Versus Deferred Cytoreductive Nephrectomy in Metastatic Renal Cell Carcinoma: A Systematic Review and Individual Patient Data Meta-analysis. Eur Urol Focus. 2025 Jan;11(1):100-108. doi: 10.1016/j.euf.2024.08.002. Epub 2024 Sep 16. PMID 39289076
- [Background] Yoshino M, Ishihara H, Nemoto Y, Nakamura K, Nishimura K, Tachibana H, Fukuda H, Toki D, Yoshida K, Kobayashi H, Iizuka J, Shimmura H, Hashimoto Y, Tanabe K, Kondo T, Takagi T. Therapeutic role of deferred cytoreductive nephrectomy in patients with metastatic renal cell carcinoma treated with nivolumab plus ipilimumab. Jpn J Clin Oncol. 2022 Oct 6;52(10):1208-1214. doi: 10.1093/jjco/hyac099. PMID 35780441
- [Background] Gross EE, Li M, Yin M, Orcutt D, Hussey D, Trott E, Holt SK, Dwyer ER, Kramer J, Oliva K, Gore JL, Schade GR, Lin DW, Tykodi SS, Hall ET, Thompson JA, Parikh A, Yang Y, Collier KA, Miah A, Mori-Vogt S, Hinkley M, Mortazavi A, Monk P, Folefac E, Clinton SK, Psutka SP. A multicenter study assessing survival in patients with metastatic renal cell carcinoma receiving immune checkpoint inhibitor therapy with and without cytoreductive nephrectomy. Urol Oncol. 2023 Jan;41(1):51.e25-51.e31. doi: 10.1016/j.urolonc.2022.08.013. Epub 2022 Oct 26. PMID 36441070
- [Background] Powles T, Blank C, Chowdhury S, Horenblas S, Peters J, Shamash J, Sarwar N, Boleti E, Sahdev A, O'Brien T, Berney D, Beltran L, Nathan P, Haanen J, Bex A. The outcome of patients treated with sunitinib prior to planned nephrectomy in metastatic clear cell renal cancer. Eur Urol. 2011 Sep;60(3):448-54. doi: 10.1016/j.eururo.2011.05.028. Epub 2011 May 17. PMID 21612860
- [Background] Bex A, Mulders P, Jewett M, Wagstaff J, van Thienen JV, Blank CU, van Velthoven R, Del Pilar Laguna M, Wood L, van Melick HHE, Aarts MJ, Lattouf JB, Powles T, de Jong Md PhD IJ, Rottey S, Tombal B, Marreaud S, Collette S, Collette L, Haanen J. Comparison of Immediate vs Deferred Cytoreductive Nephrectomy in Patients With Synchronous Metastatic Renal Cell Carcinoma Receiving Sunitinib: The SURTIME Randomized Clinical Trial. JAMA Oncol. 2019 Feb 1;5(2):164-170. doi: 10.1001/jamaoncol.2018.5543. PMID 30543350
- [Background] Mejean A, Ravaud A, Thezenas S, Colas S, Beauval JB, Bensalah K, Geoffrois L, Thiery-Vuillemin A, Cormier L, Lang H, Guy L, Gravis G, Rolland F, Linassier C, Lechevallier E, Beisland C, Aitchison M, Oudard S, Patard JJ, Theodore C, Chevreau C, Laguerre B, Hubert J, Gross-Goupil M, Bernhard JC, Albiges L, Timsit MO, Lebret T, Escudier B. Sunitinib Alone or after Nephrectomy in Metastatic Renal-Cell Carcinoma. N Engl J Med. 2018 Aug 2;379(5):417-427. doi: 10.1056/NEJMoa1803675. Epub 2018 Jun 3. PMID 29860937
- [Background] Singla N, Hutchinson RC, Ghandour RA, Freifeld Y, Fang D, Sagalowsky AI, Lotan Y, Bagrodia A, Margulis V, Hammers HJ, Woldu SL. Improved survival after cytoreductive nephrectomy for metastatic renal cell carcinoma in the contemporary immunotherapy era: An analysis of the National Cancer Database. Urol Oncol. 2020 Jun;38(6):604.e9-604.e17. doi: 10.1016/j.urolonc.2020.02.029. Epub 2020 Apr 3. PMID 32253116
- [Background] Mazzaschi G, Quaini F, Bersanelli M, Buti S. Cytoreductive nephrectomy in the era of targeted- And immuno- therapy for metastatic renal cell carcinoma: An elusive issue? A systematic review of the literature. Crit Rev Oncol Hematol. 2021 Apr;160:103293. doi: 10.1016/j.critrevonc.2021.103293. Epub 2021 Mar 2. PMID 33667661
- [Background] Zambrana F, Carril-Ajuria L, Gomez de Liano A, Martinez Chanza N, Manneh R, Castellano D, de Velasco G. Complete response and renal cell carcinoma in the immunotherapy era: The paradox of good news. Cancer Treat Rev. 2021 Sep;99:102239. doi: 10.1016/j.ctrv.2021.102239. Epub 2021 Jun 1. PMID 34157582
- [Background] Du Z, Chen W, Xia Q, Shi O, Chen Q. Trends and projections of kidney cancer incidence at the global and national levels, 1990-2030: a Bayesian age-period-cohort modeling study. Biomark Res. 2020 May 13;8:16. doi: 10.1186/s40364-020-00195-3. eCollection 2020. PMID 32435498

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT07233668/Prot_ICF_000.pdf